CLINICAL TRIAL: NCT04186637
Title: An Open-label Study of ALPN-202 in Subjects With Advanced Malignancies (NEON-1)
Brief Title: An Open-label Study of ALPN-202 in Subjects With Advanced Malignancies
Acronym: NEON-1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIS-B01
Record Dates: First submitted 2019-11-27; First posted 2019-12-05 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Advanced Solid Tumor; Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose escalation and expansion (Experimental): ALPN-202
  Interventions: Drug: ALPN-202

INTERVENTIONS:
Drug: ALPN-202 — Multiple dose levels and dose regimens of ALPN-202 will be administered

SUMMARY:
This is a cohort-based, open-label dose escalation and expansion study in adults with advanced solid tumors or lymphoma, refractory or resistant to standard therapy, or without available standard or curative therapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Adult 18 to 75 years old at screening
2. Pathologically-confirmed, locally advanced or metastatic unresectable solid tumor of an acceptable histology

   Part A (Dose Escalation)
   1. that is refractory or resistant to standard therapy, including checkpoint inhibitor(s) if approved
   2. or for which standard or curative therapy is not available

   Part B (Dose Expansion)
   1. metastatic cutaneous melanoma
   2. PD-L1-positive cancers (other than cutaneous melanoma or renal cell carcinoma)
   3. metastatic renal cell carcinoma
3. Protocol-defined measurable disease
4. Available tumor biopsy representative of current disease
5. ECOG performance status grade 0-2
6. Life expectancy of ≥ 3 months
7. Recovery to ≤ Grade 1 for any non-laboratory toxicity resulting from previous anticancer therapy prior to first dose of ALPN-202 (except alopecia, hearing loss, ≤ Grade 2 neuropathy or endocrinopathy managed with replacement therapy)
8. Adequate baseline hematologic, renal, and hepatic function

Key Exclusion Criteria:

1. History of ≥ Grade 3 immune-related adverse event leading to treatment discontinuation
2. Active or prior pneumonitis or interstitial lung disease
3. Presence of any active central nervous system metastases
4. Prior organ allograft or allogeneic hematopoietic stem cell transplantation
5. Any serious or uncontrolled health condition, which, in the opinion of the Investigator, would place the subject at undue risk from the study, impair the ability of the subject to receive protocol specified therapy, or interfere with the interpretation of study results.
6. Receipt of any protocol-restricted therapy within the timeframes indicated:

   1. PD-L1 inhibitors: 5 half-lives (e.g., atezolizumab, 135 days; avelumab, 31 days; durvalumab, 85 days)
   2. Chemotherapy, small molecule anticancer agents (e.g., kinase inhibitors), or radiation: 2 weeks
   3. Other monoclonal antibodies, antibody-drug conjugates, bispecific antibodies, antibody like drugs, cytokines, cell therapies, or radioimmunoconjugates: 4 weeks
7. Any active, known, or suspected autoimmune disease
8. Systemic treatment with corticosteroids (> 10 mg/day prednisone) or other immunosuppressive medication
9. Any second malignancy active within the previous 3 years
10. Active infection requiring therapy at the time of the first dose of ALPN-202.
11. Known seropositivity for or active infection by human immunodeficiency virus, hepatitis B or C.
12. Known allergies, hypersensitivity, or intolerance to ALPN-202 or excipients in the drug product formulation.
13. History of Grade 4 infusion-related, anaphylactic or allergic reaction to any previous Fc-based protein therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 30 days after last dose of study drug
  Type, incidence, and severity of adverse events as assessed by CTCAE

SECONDARY OUTCOMES:
Objective response | Up to 30 days after last dose of study drug
  Best observed objective responses as assessed by RECIST for solid tumors, or Lugano for lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Allison Naumovski, Ph.D., Study Director — Alpine Immune Sciences, Inc.
Locations (10):
- United States (7):
  - Investigational Site (004), Scottsdale, Arizona
  - Investigational Site (003), New Haven, Connecticut
  - Investigational Site (007), Lafayette, Indiana
  - Investigational Site (006), Louisville, Kentucky
  - Investigational Site (001), Grand Rapids, Michigan
  - Investigational Site (009), Portland, Oregon
  - Investigational Site (008), Pittsburgh, Pennsylvania
- Australia (3):
  - Investigational Site (102), Perth, Nedlands
  - Investigational Site (101), Melbourne, Victoria
  - Investigational Site (103), Melbourne, Victoria

REFERENCES:
- [Derived] Davar D, Cavalcante L, Lakhani N, Moser J, Millward M, McKean M, Voskoboynik M, Sanborn RE, Grewal JS, Narayan A, Patnaik A, Gainor JF, Sznol M, Enstrom A, Blanchfield L, LeBlanc H, Thomas H, Chisamore MJ, Peng SL, Naumovski A. Phase I studies of davoceticept (ALPN-202), a PD-L1-dependent CD28 co-stimulator and dual PD-L1/CTLA-4 inhibitor, as monotherapy and in combination with pembrolizumab in advanced solid tumors (NEON-1 and NEON-2). J Immunother Cancer. 2024 Aug 3;12(8):e009474. doi: 10.1136/jitc-2024-009474. PMID 39097413